CLINICAL TRIAL: NCT01426971
Title: National, Controlled, Randomized, Double-blind, Parallel Study to Investigate the Efficacy of 2 Capsules of Ibuprofen 400mg in Association With Caffeine 100mg in Fixed Dose Combination Compared to Two Capsules of Ibuprofen 400mg in the Treatment of Migraine
Brief Title: Ibuprofen Versus Ibuprofen Plus Caffeine in the Treatment of Migraine.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBUCA_L_05619
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Pain
Keywords: Migraine
MeSH Terms: conditions — Pain; Migraine Disorders | interventions — Ibuprofen; Caffeine

ARMS (2):
- Ibuprofen+caffeine (Experimental): 2 capsules
  Interventions: Drug: IBUPROFEN + CAFFEINE
- Ibuprofen (Active Comparator): 2 capsules
  Interventions: Drug: IBUPROFEN

INTERVENTIONS:
Drug: IBUPROFEN + CAFFEINE — Pharmaceutical form: capsule Route of administration: oral
  Arms: Ibuprofen+caffeine
Drug: IBUPROFEN — Pharmaceutical form: capsule Route of administration: oral
  Arms: Ibuprofen

SUMMARY:
Primary Objective:

- To compare the treatment groups in the reduction of pain score by at least 30 mm on a visual pain scale (VAS) at 60 minutes after study medication intake, compared to the baseline score (obtained before the study medication intake).

Secondary Objectives:

* To assess the proportion of patients with more than 50% pain relief, according to the VAS score at 45 minutes after study medication intake compared to baseline
* Determine the following aspects in the timing of study medication intake:

  * Time to the first perception of pain relief
  * Time to onset of meaningful pain relief
  * Reduction of pain at 15, 30, 45, 60, 120 and 240 minutes after study medication intake, to be evaluated as the difference between the scores on VAS in each period and baseline
* To assess the pain according to the five items of Headache Relief Rating - HRR (0: strong worsening 1: slight worsening 2: no change 3: slight improvement 4: strong improvement) at 15, 30, 45 and 60 minutes after study medication intake, according to the diaries completed by the patients
* To check the proportion of the patients requiring the third tablet of study medication within 24 hours of starting the study treatment and when it occurred
* To check the timing and frequency of rescue medication intake, as well as the proportion of patients who used these medications within 24 hours of starting the treatment
* Safety assessment.

ELIGIBILITY:
Inclusion criteria:

* 18 years old to less ore equal than 65 with migraine defined according to the criteria of the headache Classification Committee (ICHD II) of the International Headache Society (HIS)
* Migraine first onset before 50 years old
* Occurrence of at least one episode every two months or up to 8 episodes per month during the previous 3 months, which must not exceed 14 days per month
* Pain relief with the use of Over The Counter (OTC) medicines by at least 75% of episodes
* Headache of at least moderate intensity (VAS greater than 30 mm), at least 75% of episodes
* Absence of caffeine and black tea at least 2 hours before and one hour after drug administration

Exclusion criteria:

* Use of acupuncture, homeopathy and/or phytotherapy
* Use of Tryptanes in the last 30 hours, no steroidal anti-inflammatory drugs in the last 48 hours and analgesics in the last 15 hours
* Use of analgesics drug products for more than 10 days per month, consecutive or not, for a period exceeding three months
* Other types of headache that is not migraine, according to the International Classification of Headache Disorders (ICHD II)
* Chronic and complicated migraine, according to ICHD II
* Coexisting disease or significant medical conditions which in the investigators judgment interfere and/or prevent the individuals proper participation in the study
* Treatment with methotrexate, glucocorticoids, anticoagulants and/or lithium
* Hypersensibility to study medication (or any component of the formula), to acetyl salicylic, no steroidal anti-inflammatory drugs and/or any other analgesic or antipyretic
* Nasal polyps, asthma and / or other allergic manifestations
* Subjects with edema, diarrhea and/or vomiting, who are not eating or drinking fluids properly according to the investigators judgment or experiencing visual disorders
* Use of antihypertensive medications and/or psychoactive in the last 6 months
* History of anorexia, bulimia and/or mental disorders
* History of tachycardia, arrhythmia, congestive heart failure, coronary artery disease and/or coagulopathy
* History of thyroid disease and/or parathyroid disease, liver disease and/or gastrointestinal
* History of dyspeptic disorder, including gastritis, peptic ulcer and/or gastrointestinal bleeding
* Impaired renal function tests and/or history of renal disease, including kidney failure
* Pregnant (or planning to become pregnant during the course of the study) or who are breast feeding
* Woman in childbearing age, childbearing potential not protected by an effective contraceptive method of birth control. Status of pregnancy should be checked for pregnancy test serum or urine before exposure to the Investigational product.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with reduction of at least 30mm in the visual scale (VAS) of pain | from baseline to 60 minutes

SECONDARY OUTCOMES:
Number of patients with more than 50% of pain reduction | up to 45 minutes
Median time of the first perception of pain relief since study medication intake | 4 hours
Median time to onset of significant pain relief compared to the time of study medication intake | 4 hours
Headache Relief Rating score (HRR) | up to 60 mins
Mean of VAS difference between each time after medication intake and the baseline. | 15, 30, 45, 60, 120 and 240 minutes post dose
Number of patients who used the third tablet of study medication | up to 24 hours
Number of patients requiring rescue medication | up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi